CLINICAL TRIAL: NCT04266548
Title: Superselective Intra-arterial Hepatic Injection of Indocyanine Green (ICG) for Fluorescence Image-guided Segmental Positive Staining
Brief Title: Arterial Base Fluorescence Segmental Positive Staining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGMH-20170147A3
Record Dates: First submitted 2020-02-06; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Hepatic Carcinoma
Keywords: indocynide green; Image guide surgery; near infra-red laparoscopy; laparoscopic hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: The study was the clinical feasibility study. Only selected single HCC patients was enrolled to study the feasibility of image guide surgery for laparoscopic hepatectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- super-selective hepatic artery ICG injection group (Experimental): single arm for feasibility study of intra-hepatic artery base fluorescent segmental demarcation
  Interventions: Procedure: Superselective Intra-arterial Hepatic Injection of Indocyanine Green (ICG) for Fluorescence Image-guided Segmental Positive Staining

INTERVENTIONS:
Procedure: Superselective Intra-arterial Hepatic Injection of Indocyanine Green (ICG) for Fluorescence Image-guided Segmental Positive Staining — The patients with single HCC which is planned to received laparoscopic hepatectomy were involved. Procedures were performed in conventional angiography room. The celiac trunk was catheterized and a microcatheter was advanced into segmental hepatic artery branches which supplied the HCC. The 5cc 0.125 mg/cc ICG was injected from super-selective hepatic artery in operative room. A Near-Infrared laparoscope was used to detect the fluorescent signal to assess the correspondence between arterial-based fluorescence demarcation and ultrasound-based surgical demarcation.

SUMMARY:
More and more laparoscopic hepatectomy were performed due to increasing experience, well designed instruments and energy device. But the localization of tumor and resection line design are still relative difficult comparing open approach due to limit space. Intraoperative liver segmentation can be obtained by ultrasound-guide intraportal injection of a fluorophore and illuminating with a Near-Infrared light source for positive staining and by intravenous injection after ligation of segmental vessels for negative staining .The ultrasound guide intraportal injection approach is challenging in the minimally-invasive setting. However hepatocelluar carcinoma(HCC) was supplied by hepatic artery mainly. The investigators aimed to evaluate the feasibility of arterial base positive staining for fluorescence liver segmentation in human by superselective intra-hepatic artery injection of Indocyanine Green (ICG) .

DETAILED DESCRIPTION:
Materials and Methods

1. Participants The present prospective, single-center, feasibility study of fluorescence demarcation of hepatic segment including HCC by means of direct super-selective intrahepatic artery ICG injection. Patients were enrolled according to the following criteria: single HCC, scheduled for laparoscopic hepatectomy for curative resection, age ranging from 20 to 85 years old, absence of proven or suspected allergies to iodine or ICG, absence of coagulopathy, absence of diseases contraindicating general anesthesia, and absence of pregnancy.

   All the bio-chemical test, cardiac echo , cardiac thalium test, ICG clearance test, Liver CT or MRI were obtained before operation
2. Equipment Endovascular procedure was performed in the conventional angiography room and laparoscopic hepatecotmy was done in operating room at the Kaohsiung Chang Gung memorial hospital. Near infra-red fluorescence laparoscopy was used to acquire the fluorescence signal arising from the liver parenchyma after Indocyanine Green (ICG) injection.
3. Procedures

   1. Celiac trunk angiography and super-selective hepatic angiography:

      A 4 Fr angiography sheath (Terumo Europe NV, Belgium) was placed under aseptic conditions in the right femoral artery, using the Seldinger technique. A 4 Fr Cobra-2 catheter (Terumo Europe NV, Belgium) was positioned at the origin of the celiac trunk. A selective celiac trunk digital subtraction angiographic (DSA) run was performed, after injection of a contrast medium (Visipaque 270, GE Healthcare; Buckinghamshire, United Kingdom), 28mL at a rate of 4mL/sec. A 2.7 French micro-catheter (Progreat™, Terumo Europe NV; Belgium) was used to super-selectively catheterize different hepatic segmental arteries supplying the target hepatic segment including HCC. In all cases, the position was controlled by performing DSA and angio computer tomography runs with selective micro-catheter injections. The micro-catheter was then perfused with saline and left in place until surgery. Then the patients were transferred to operative room while operative room available.
   2. Evaluation of hepatic segmental demarcation using NIR real-time imaging during laparoscopic hepatectomy:

The patients underwent a standard 5-port laparoscopic hepatectomy, which was performed by 2 experienced laparoscopic surgeons .

Stage I : the liver mobilization was performed for preparing the hepatectomy. The intraoperative ultrasound was used for localization of HCC. The resection line was defined as principle of laparoscopic hepatectomy such as surgical margin, surgical volume and etc. The pringle control device was prepared.

Stage II : Rea-time enhanced visualization of the hepatic segment which were supplied feeding artery was achieved by means of fluorescence imaging using a direct selective intrahepatic artery injection of a 5 mL bolus of ICG (DiagnoGreen®, Taiwan, ROC) at a concentration of 0.125mg/mL. The demarcation of enhanced hepatic segment were defined. The correspondence between the fluorescence margin and ultrasound(US) guide resection line were analized.

Stage III: The surgical resection line was chose by real time clinical judgement including analysis of information of US, artery-base CT, fluorescence image, liver anatomy and patient condition. The laparoscopic hepatectomy was performed with pringle vascular control.

Stage IV: the specimen information including tumor size and margin in vitro was recoded. The distance between surgical margin and enhanced liver were measured.

ELIGIBILITY:
Inclusion Criteria:

* Single Hepatocellular carcinoma.
* plan of Laparoscopic hepatectomy.
* Age between 20 to 85 y/o.

Exclusion Criteria:

* allergies to iodine or ICG
* Liver cirrhosis
* coagulopathy
* chronic kidney disease
* pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Fluorescent hepatic segment demarcation area | intra-operative period
  The surface size of fluorescent enhanced hepatic segment were measured as cm x cm .
the rate of fluorescent demarcation corresponding to US guide resection area | intra-operative period
  The evaluation of the fluorescent hepatic surface which is included in the resected area or not
The minimal distance between tumor and fluorescent margin | intra-operative period
  The distance between tumor edge and fluorescent parenchyma edge was measured as cm. This purpose was to evaluation the oncologic safety if the resection line is following the fluorescent margin
The minimal surgical margin | intra-operative period
  The distance between tumor edge and resected parenchyma edge was measured as cm.
surgical benefit rate of fluorescent image | intra-operative period
  If the fluorescent enhanced area is similar to resected parenchyma or the information of fluorescent image change the primary surgical plan, it was indicated benefit for surgery.

SECONDARY OUTCOMES:
Post operative complication | one months after operation
  any complication related to surgery
Post operative angiography procedure complication | one months after operation
  any complication related to angiography procedure
Post operative hospital stay | one months after operation
  The day in hospital after operation
Post operative Mortality | any complication related to surgery
  any mortality related to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Yin Liu, MD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Niaosong, Kaohsiung, Taiwan

IPD SHARING:
Plan to Share IPD: No
due to special technique, data is unique and difficult to fit with other study

REFERENCES:
- [Background] Diana M, Liu YY, Pop R, Kong SH, Legner A, Beaujeux R, Pessaux P, Soler L, Mutter D, Dallemagne B, Marescaux J. Superselective intra-arterial hepatic injection of indocyanine green (ICG) for fluorescence image-guided segmental positive staining: experimental proof of the concept. Surg Endosc. 2017 Mar;31(3):1451-1460. doi: 10.1007/s00464-016-5136-y. Epub 2016 Aug 5. PMID 27495341
- [Result] Ishizawa T, Gumbs AA, Kokudo N, Gayet B. Laparoscopic segmentectomy of the liver: from segment I to VIII. Ann Surg. 2012 Dec;256(6):959-64. doi: 10.1097/SLA.0b013e31825ffed3. PMID 22968066
- [Result] Ferrero A, Lo Tesoriere R, Russolillo N, Vigano L, Forchino F, Capussotti L. Ultrasound-guided laparoscopic liver resections. Surg Endosc. 2015 Apr;29(4):1002-5. doi: 10.1007/s00464-014-3762-9. Epub 2014 Aug 19. PMID 25135446
- [Result] Shindoh J, Seyama Y, Matsuda M, Miyata Y, Shida D, Maeshiro T, Miyamoto S, Inoue S, Umekita N. Continuous ultrasound navigation for safe and precise anatomic resection of the liver. Hepatogastroenterology. 2013 May;60(123):590-4. doi: 10.5754/hge12861. PMID 23282740
- [Result] Rethy A, Lango T, Marvik R. Laparoscopic ultrasound for hepatocellular carcinoma and colorectal liver metastasis: an overview. Surg Laparosc Endosc Percutan Tech. 2013 Apr;23(2):135-44. doi: 10.1097/SLE.0b013e31828a0b9a. PMID 23579506
- [Result] Makuuchi M, Hasegawa H, Yamazaki S. Ultrasonically guided subsegmentectomy. Surg Gynecol Obstet. 1985 Oct;161(4):346-50. PMID 2996162
- [Result] Gotoh K, Yamada T, Ishikawa O, Takahashi H, Eguchi H, Yano M, Ohigashi H, Tomita Y, Miyamoto Y, Imaoka S. A novel image-guided surgery of hepatocellular carcinoma by indocyanine green fluorescence imaging navigation. J Surg Oncol. 2009 Jul 1;100(1):75-9. doi: 10.1002/jso.21272. PMID 19301311
- [Result] Tanaka T, Takatsuki M, Hidaka M, Hara T, Muraoka I, Soyama A, Adachi T, Kuroki T, Eguchi S. Is a fluorescence navigation system with indocyanine green effective enough to detect liver malignancies? J Hepatobiliary Pancreat Sci. 2014 Mar;21(3):199-204. doi: 10.1002/jhbp.17. Epub 2013 Jul 1. PMID 23818301
- [Result] Aoki T, Yasuda D, Shimizu Y, Odaira M, Niiya T, Kusano T, Mitamura K, Hayashi K, Murai N, Koizumi T, Kato H, Enami Y, Miwa M, Kusano M. Image-guided liver mapping using fluorescence navigation system with indocyanine green for anatomical hepatic resection. World J Surg. 2008 Aug;32(8):1763-7. doi: 10.1007/s00268-008-9620-y. PMID 18543027
- [Result] Ishizawa T, Zuker NB, Kokudo N, Gayet B. Positive and negative staining of hepatic segments by use of fluorescent imaging techniques during laparoscopic hepatectomy. Arch Surg. 2012 Apr;147(4):393-4. doi: 10.1001/archsurg.2012.59. No abstract available. PMID 22508790
- [Result] Sakoda M, Ueno S, Iino S, Hiwatashi K, Minami K, Kawasaki Y, Kurahara H, Mataki Y, Maemura K, Uenosono Y, Shinchi H, Natsugoe S. Anatomical laparoscopic hepatectomy for hepatocellular carcinoma using indocyanine green fluorescence imaging. J Laparoendosc Adv Surg Tech A. 2014 Dec;24(12):878-82. doi: 10.1089/lap.2014.0243. PMID 25347551
- [Derived] Li WF, Al-Taher M, Yu CY, Liu YW, Liu YY, Marescaux J, Cheng YF, Diana M, Wang CC. Super-Selective Intra-Arterial Indocyanine Green Administration for Near-Infrared Fluorescence-Based Positive Staining of Hepatic Segmentation: A Feasibility Study. Surg Innov. 2021 Dec;28(6):669-678. doi: 10.1177/1553350621996972. Epub 2021 Mar 31. PMID 33787401